CLINICAL TRIAL: NCT04927793
Title: A Phase I, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]EDP-938 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Absorption, Metabolism, and Excretion (AME) Study of [14C]EDP-938 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 938-009
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: AME Study
MeSH Terms: interventions — EDP-938

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm EDP-938 (Experimental)
  Interventions: Drug: EDP-938

INTERVENTIONS:
Drug: EDP-938 — [14C]EDP-938

SUMMARY:
A Phase 1, Open-label Study of the absorption, metabolism, and excretion of a single oral dose of [14C]EDP-938 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males of any ethnic origin, between 18 and 55 years of age, inclusive.
* Able to comprehend and willing to sign an Informed Consent Form
* In good health, determined by no clinically significant findings from medical history, physical examination (check-in only), 12-lead ECG, vital signs measurements, and clinical laboratory evaluations

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of stomach or intestinal surgery or resection, including cholecystectomy, that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).

  a. Subjects with a history of cholecystitis, cholelithiasis, and/or choledocholithiasis will also be excluded.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* A body surface area-adjusted estimated glomerular filtration rate (eGFR) ≤ 90 mL/min per 1.73 m2 according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-938 in plasma | Up to 11 days
AUC0-tlast of EDP-938 in plasma | Up to 11 days
AUC-inf in plasma | Up to 11 days
Amount excreted in urine (Aeu) | Up to 11 days
Amount excreted in feces (Aef) | Up to 11 days
Cmax of EDP-938 metabolites in plasma | Up to 11 days

SECONDARY OUTCOMES:
Safety measured by occurrence of adverse events | Up to 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No